CLINICAL TRIAL: NCT01356290
Title: A Phase II Study of Metronomic and Targeted Anti-angiogenesis Therapy for Children with Recurrent/progressive Medulloblastoma, Ependymoma and ATRT
Brief Title: Antiangiogenic Therapy for Children with Recurrent Medulloblastoma, Ependymoma and ATRT
Acronym: MEMMAT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Andreas Peyrl, MD, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MUV-MEMMAT-01
Record Dates: First submitted 2011-05-17; First posted 2011-05-19 (Estimated); Last update posted 2024-10-21 (Actual); Status verified 2024-01

CONDITIONS: Medulloblastoma Recurrent; Ependymoma Recurrent; ATRT Recurrent
Keywords: Medulloblastoma; Ependymoma; ATRT; Relapse; Children; antiangiogenic; metronomic; intraventricular
MeSH Terms: conditions — Medulloblastoma; Ependymoma; Recurrence | interventions — Bevacizumab; Thalidomide; Celecoxib; fenofibric acid; Etoposide; Cyclophosphamide; etoposide phosphate; Cytarabine

STUDY DESIGN:
Intervention Model Description: 3 Strata (medulloblastoma - 40 patients; ependymoma - 30 patients; ATRT - 30 patients)
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Bevacizumab — 10mg/kg, intravenous (iv), biweekly, 1 year
  Other Names: Avastin
Drug: Thalidomide — 3mg/kg, oral, daily, 1 year
Drug: Celecoxib — 50-400mg, oral bid, daily, 1 year
Drug: Fenofibric acid — 90mg/m2, oral, daily, 1 year
Drug: Etoposide — 35-50 mg/m2, oral, alternating 21-day cycles of daily oral etoposide and cyclophosphamide, 1 year
Drug: Cyclophosphamide — 2.5mg/kg, oral, alternating 21-day cycles of daily oral etoposide and cyclophosphamide, 1 year
Drug: Etoposide phosphate — 0.5mg, intrathecal, day 1-5, every four weeks, alternating with intrathecal liposomal cytarabine, 1 year
Drug: Cytarabine — 16-30mg, intrathecal, twice weekly for two weeks out of every four weeks, alternating with intrathecal etoposide phosphate, 1 year

SUMMARY:
Patients with relapsed medulloblastoma, ependymoma and ATRT have a very poor prognosis whether treated with conventional chemotherapy, high-dose chemotherapy with stem cell rescue, irradiation or combinations of these modalities. Antiangiogenetic therapy has emerged as new treatment option in solid malignancies. The frequent, metronomic schedule targets both proliferating tumor cells and endothelial cells, and minimizes toxicity. In this study the investigators will evaluate the use of biweekly intravenous bevacizumab in combination with five oral drugs (thalidomide, celecoxib, fenofibrate, and alternating cycles of daily low-dose oral etoposide and cyclophosphamide), augmented with alternating courses of intrathecal etoposide and cytarabine. The aim of the study is to extend therapy options for children with recurrent or progressive medulloblastoma, ependymoma and ATRT, for whom no known curative therapy exists, by prolonging survival while maintaining good quality of life. The primary objective of the MEMMAT trial is to evaluate the activity of this multidrug antiangiogenic approach in these heavily pretreated children and young adults. Additionally, progression-free survival (PFS), overall survival (OS), as well as feasibility and toxicity will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or progressive medulloblastoma, ependymoma or ATRT (at least one site of untreated recurrent disease)
* Histological confirmation of medulloblastoma, ependymoma or ATRT at diagnosis or relapse
* Female or male, aged from 0 to <20 years (at time of original diagnosis)
* Participants must have normal organ and bone marrow function (ALT <5x institutional upper limit of normal, creatinine <1.5x institutional upper limit of normal for age, WBC >1000/mm3, platelets > 20,000/mm3. Patients with values less than WBC 2000/mm3 or platelets 50,000/mm3 will require initiation of treatment with etoposide and cyclophosphamide at a lower starting dose as defined within the protocol.
* Karnofsky performance status ≥50. For infants and children less than 12 years of age, the Lansky play scale ≥50% will be used
* Written informed consent of patients and / or parents

Exclusion Criteria:

* Active infection
* VP-shunt dependency
* Pregnancy or breast feeding
* Conventional chemotherapy, antiangiogenic treatment or complete irradiation of all disease for current relapse (surgery may be performed before antiangiogenic treatment; patients with sites of disease not irradiated are still eligible for the protocol)
* Known hypersensitivity to any of the drugs in the protocol
* Active peptic ulcer
* Any significant cardiovascular disease not controled by standard therapy e.g. systemic hypertension
* Anticipation of the need for major elective surgery during the course of the study treatment
* Any disease or condition that contraindicates the use of the study medication/treatment or places the patient at an unacceptable risk of experiencing treatment-related complications
* Non-healing surgical wound
* A bone fracture that has not satisfactorily healed

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 8 years
  Response rate (Complete remission, partial response, stable disease =[CR+PR+SD]/n) 6 months after start of antiangiogenic treatment

SECONDARY OUTCOMES:
Overall survival rate | 8 years
  The percentage of patients in the study who are alive for a certain period of time (6, 12, 24, and 36 months) after start of treatment with an antiangiogenic multidrug-regime
Progression free survival rate | 8 years
  The percentage of patients in the study who are alive with a non-progressive disease for a certain period of time (6, 12, 24, and 36 months) after start of treatment with an antiangiogenic multidrug-regime.
Toxicity | 8 years
  To evaluate and document toxicities from chronic administration of these drugs at the doses prescribed in this protocol in patients with recurrent or progressive medulloblastoma. These will be descriptive in nature.
Feasibility | 6 years
  To evaluate the feasibility of achieving the prescribed drug doses given the reduced bone marrow tolerance after multiple relapses.
Quality of life | 8 years
  Quality of Life (QoL) will be evaluated by a generic quality of life instrument for children (the KINDL®-questionnaire).
Prognostic factors | 8 years
  To evaluate the influence of tumor biology(histologic subgroups, metastatic stage, age at first diagnosis [<3 years, >3 years]), age at start of antiangiogenic therapy, sex, duration of remission prior to antiangiogenic therapy, number of recurrences.
Angiogenic factors | 8 years
  To evaluate serum markers for in-vitro correlative studies of tumor response.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Peyrl, MD, Principal Investigator — Medical University of Vienna; Monika Chocholous, MD, Study Chair — Medical University of Vienna
Locations (22):
- United States (4):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute and Boston Children's Hospital, Boston, Massachusetts
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Dell Children's Medical Group SFC-HEM/ONC, Austin, Texas
- Austria (5):
  - Medical University of Graz, Graz
  - Medical University of Innsbruck, Innsbruck
  - Kepler Universitätsklinikum Med Campus IV, Linz
  - Salzburger Universitätsklinikum, Salzburg
  - Medical University of Vienna, Vienna
- Czechia (2):
  - University Hospital Brno, Brno
  - Motol University Hospital Prague, Prague
- University hospital Rigshospitalet, Copenhagen, Denmark
- France (2):
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
- Onkologisk-hematologisk seksjon Barneklinikken Haukeland universitetssjukehus, Bergen, Bergen, Norway
- Hospital Infantil Universitario Nino Jesus, Madrid, Spain
- Sweden (6):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Universitetssjukhuset Linköping, Linköping
  - Skånes universitetssjukhus, Lund
  - Karolinska University Hospital, Stockholm
  - Norrlands Universitetssjukhus, Umeå
  - Akademiska sjukhuset, Uppsala

REFERENCES:
- [Derived] Peyrl A, Chocholous M, Sabel M, Lassaletta A, Sterba J, Leblond P, Nysom K, Torsvik I, Chi SN, Perwein T, Jones N, Holm S, Nyman P, Morse H, Oberg A, Weiler-Wichtl L, Leiss U, Haberler C, Schmook MT, Mayr L, Dieckmann K, Kool M, Gojo J, Azizi AA, Andre N, Kieran M, Slavc I. Sustained Survival Benefit in Recurrent Medulloblastoma by a Metronomic Antiangiogenic Regimen: A Nonrandomized Controlled Trial. JAMA Oncol. 2023 Dec 1;9(12):1688-1695. doi: 10.1001/jamaoncol.2023.4437. PMID 37883081
- [Derived] Slavc I, Mayr L, Stepien N, Gojo J, Aliotti Lippolis M, Azizi AA, Chocholous M, Baumgartner A, Hedrich CS, Holm S, Sehested A, Leblond P, Dieckmann K, Haberler C, Czech T, Kool M, Peyrl A. Improved Long-Term Survival of Patients with Recurrent Medulloblastoma Treated with a "MEMMAT-like" Metronomic Antiangiogenic Approach. Cancers (Basel). 2022 Oct 19;14(20):5128. doi: 10.3390/cancers14205128. PMID 36291912